CLINICAL TRIAL: NCT00416013
Title: Correlations Between BNP and Dry Weight, and Between Troponin and Mortality, in Hemodialysis Patients
Brief Title: Correlations Between BNP & Dry Weight, and Between Troponin & Mortality, in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Abbott RDx Cardiometabolic (Other)
Responsible Party: Mark Flemmer, MD, Eastern Virginia Medical School
Other Study IDs: EVMS 05-08-EX-0246
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Kidney Failure, Chronic; Heart Failure, Congestive
Keywords: Beta Natriuretic Peptide; Troponin; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Beta Natriuretic Peptide (BNP) is regarded as the most sensitive test for congestive heart failure (CHF). BNP has also been found to be highly predictive of other conditions including pulmonary hypertension, pulmonary embolism and in the general population where mild increases are associated with stroke and heart attack. BNP is also weakly and variably correlated with renal function.

We believe that each dialysis patient will have an ideal or "dry" BNP level which will accurately and reproducibly reflect their optimal fluid status. Secondary hypotheses are that baseline BNP and troponin, as well as changes in BNP and troponin during dialysis, will be highly predictive of mortality and adequacy of dialysis.

DETAILED DESCRIPTION:
Plasma BNP is regarded as the most sensitive test for congestive heart failure (CHF). Multiple studies have shown that BNP is a distress hormone released by the distended left ventricular myocardium which correlates significantly with left ventricular wedge pressure and all-cause mortality in those with CHF and acute coronary syndromes. BNP has also been found to be highly prognostic across a wide variety of other conditions including pulmonary hypertension, pulmonary embolism and in the general population where mild increases are associated with stroke and heart attack. BNP is weakly and variably correlated with renal function. How much of this elevation is related to renal clearance or the perturbations of the circulation that uremia, hypertension and chronic fluid overload cause is speculative.

There is a paucity of information about BNP levels in hemodialysis (HD) patients. Intuitively, BNP levels should be an ideal marker for left ventricular preload or dry weight in the HD population. Furthermore since BNP has a short half-life of 20 minutes, serial measurements during dialysis would be expected to rapidly reflect ultrafiltration and fluid status. Currently the amount of fluid removed during dialysis is defined clinically by inter-dialysis weight gain, hypertension, edema or dyspnea. Accurate assessment of ideal or dry weight is critically important in HD patients as both fluid overload and intravascular dehydration can have fatal consequences in this very frail population.

The few published articles on BNP as a marker for adequacy of dialysis have given conflicting data and have been flawed by both small sample size and not doing sequential measurements on each patient.

Cardiac troponins are well-established markers of myocardial injury. Both troponin I and T subtypes are regulatory proteins that help coordinate the actions of actin and myosin. Existing both in the cytosol and in the structure of the myocardium, their release is believed to correlate with the breakdown of actin and myosin in the area of myocardial damage. Elevated troponin levels have also been correlated with pulmonary embolism and other sources of right heart strain. Their use in the setting of patients with ESRD has been less clear. Sampling of asymptomatic ESRD patients found a significant percentage of them to have elevated troponins. Proposed mechanisms for this increase include impaired renal excretion, left ventricular hypertrophy, endothelial dysfunction, stretch mediated troponin release, and leakage of cytoplasmic free troponin secondary to poor membrane integrity. Regardless of the mechanism, a large study of asymptomatic patients found significantly increased mortality in those with increased troponins.

While the correlation between increased troponins and mortality has been shown, the effects of hemodialysis on troponin levels has yet to be demonstrated in published studies.

HYPOTHESIS: We believe that each dialysis patient will have an ideal or "dry" BNP level which will accurately and reproducibly reflect their optimal fluid status. Subsidiary hypotheses are that baseline BNP and troponin, as well as changes in BNP and troponin during dialysis, will be highly predictive of mortality and adequacy of dialysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients who complete dialysis, are 18 years or older or 85 years or less, and give informed consent will be eligible.

Exclusion Criteria:

* Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End Stage Renal Disease (ESRD) patients on hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2005-12; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Flemmer, MBB Ch, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States